CLINICAL TRIAL: NCT00076570
Title: Depletion Induction With Rabbit Anti-Thymocyte Globulin, Followed by Two Approaches Toward Monotherapy Immunosuppression in Kidney Transplant Recipients
Brief Title: Combination Drug Therapy Followed by Single Drug Steroid Free Therapy to Prevent Organ Rejection in Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040099; 04-DK-0099
Record Dates: First submitted 2004-01-26; First posted 2004-01-27 (Estimated); Results first posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-08

CONDITIONS: Kidney Transplantation
Keywords: Tolerance; Kidney; Transplant; Polyclonal; Antibody; Kidney Transplant
MeSH Terms: interventions — Sirolimus; Tacrolimus

ARMS (2):
- Sirolimus (Experimental): Patients are treated with combination therapy with both sirolimus and tacrolimus for 6 month. After 6 months, patients are switched to sirolimus monotherapy and followed up for 4 years.
  Interventions: Drug: Sirolimus
- Tacrolimus (Active Comparator): Patients are treated with combination therapy with both sirolimus and tacrolimus for 6 month. After 6 months, patients are switched to tacrolimus monotherapy and followed up for 4 years.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Sirolimus
  Arms: Sirolimus
Drug: Tacrolimus
  Arms: Tacrolimus

SUMMARY:
This study will test the safety and effectiveness of a combination of three drugs followed by long-term treatment with just one drug in preventing organ rejection in kidney transplant patients. Current anti-rejection medicines are not completely effective in preventing rejection. This trial will test how well Thymoglobulin, Tacrolimus, and Sirolimus work together post-transplant and if the treatment can be reduced over time to control rejection with either Tacrolimus or Sirolimus alone.

Candidates for kidney transplantation at the National Institutes of Health Clinical Center may participate in this 5-year study. Patients will be screened for eligibility with a medical history, physical examination, and blood tests.

Participants will undergo the following tests and procedures:

* Central line placement: A large intravenous catheter (plastic tube, or IV line) is placed in a vein in the chest or neck under local anesthesia before the transplant surgery. The line remains in place for some time during the hospitalization to administer Thymoglobulin, antibiotics, and blood, if needed. The line is also used to collect blood samples.
* Leukapheresis: This procedure for collecting white blood cells is done before the transplant. The cells are studied to evaluate the patient's immune system. Whole blood is withdrawn through a catheter in an arm vein or through the central line and directed into a machine that separates the blood components by spinning. The white cells are removed and the red cells and plasma are returned to the body.
* Kidney transplant: Patients undergo kidney transplant surgery under general anesthesia.
* Immunosuppressive therapy: Patients receive thymoglobulin by vein for 4 days starting 1 day before the transplant. They also take Tylenol, Benadryl and a steroid (methylprednisolone) to help reduce the side effects of the Thymoglobulin. After the transplant, patients receive Tacrolimus and Sirolimus by mouth once a day for 6 months and then either Tacrolimus or Sirolimus alone indefinitely. In addition, they take medicines to help prevent viral and fungal infections for 6 months because the immunosuppressive therapy leaves them vulnerable to infection.
* Follow-up visits: After hospital discharge, patients return to the Clinical Center twice a week for 4 weeks, then every 6 months for 1 year, and then yearly for another 4 years. At each visit, the patient's vital signs are checked and blood and urine samples are collected. Periodically, patients are also questioned about how they feel and how the transplant has affected their quality of life. Kidney biopsies (removal of a small amount of kidney tissue through a thin needle) are done when the patient begins single-drug immunosuppression (generally 6 months after transplantation) and 1 year after that. The biopsied tissue is examined to evaluate how well the kidney is responding to the treatment and to determine how to proceed with therapy.
* Routine laboratory tests: Routine tests, coordinated by the patient's local physician, are done 2 to 3 times a week for the first 2 to 3 months after transplantation, then weekly for several more months, and at least monthly for life.

DETAILED DESCRIPTION:
This protocol facilitates the development of methods for determining whether transplant recipients have developed immune hyporesponsiveness or tolerance towards their allograft. These methods will involve the study of peripheral blood or biopsy tissue obtained at regular intervals from patients receiving kidney or combined kidney-pancreas allografts at the NIH Clinical Center. In addition, patients that have previously received a kidney or combined kidney-pancreas allograft will be evaluated using assays requiring peripheral blood mononuclear cells and/or biopsies. Assays developed under this protocol will be used in subsequent protocols to assess the effects of immune modulating treatment regimens and may eventually be used to direct clinical care or guide the withdrawal of immunosuppressive agents. However, patients enrolled in this protocol will not have any change in treatment based solely on the assays developed without being enrolled in an additional study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Candidates for a kidney transplant at the Clinical Center.

Willingness and legal ability to give informed consent.

Availability of donor tissue for testing. This could include splenic or peripheral blood lymphocytes from a cadaveric donor or a willing living donor who consents to periodic phlebotomy for peripheral blood lymphocyte isolation.

EXCLUSION CRITERIA:

Immunosuppressive drug therapy at the time of or 2 months prior to enrollment. Specifically, candidates may not be taking prednisone, cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, anti-lymphocyte agents, cyclophosphamide, methotrexate, or other agents whose therapeutic effect is immunosuppressive.

Any active malignancy or any history of any hematogenous malignancy or lymphoma. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing the lesions are appropriately treated prior to transplant.

Any known immunodeficiency syndrome, or other condition that, in the opinion of the investigators, would likely increase the risk of protocol participation or confound the interpretation of the data.

Any history of sensitization to rabbits or extensive exposure to rabbits, as defined by symptomatic allergic response upon exposure to rabbits.

Inability or unwillingness to comply with protocol monitoring and therapy including, among others, a history of noncompliance, circumstances where compliance with protocol requirements is not feasible due to living conditions, travel restrictions, access to urgent medical services, or access to anti-rejection drugs after the research protocol is completed.

Peak Panel Reactive Antibody greater than 20%, or historically positive crossmatch due to HLA (human leukocyte antigen)-specific antibodies.

HLA (human leukocyte antigen) identity between the donor and recipient.

Pregnancy or unwillingness to practice an approved method of birth control. Acceptable methods of birth control may include barrier methods (condom and/or diaphragm with spermicide), oral contraceptives, Norplant, Depo-Provera or partner sterility.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique E Cho, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Eggers PW. Effect of transplantation on the Medicare end-stage renal disease program. N Engl J Med. 1988 Jan 28;318(4):223-9. doi: 10.1056/NEJM198801283180406. PMID 3275896
- [Background] Hariharan S, Johnson CP, Bresnahan BA, Taranto SE, McIntosh MJ, Stablein D. Improved graft survival after renal transplantation in the United States, 1988 to 1996. N Engl J Med. 2000 Mar 2;342(9):605-12. doi: 10.1056/NEJM200003023420901. PMID 10699159
- [Background] Barry JM. Immunosuppressive drugs in renal transplantation. A review of the regimens. Drugs. 1992 Oct;44(4):554-66. doi: 10.2165/00003495-199244040-00003. PMID 1281071
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-DK-0099.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Totally 31 patients were enrolled during August 2002 to October 2006 at NIH clinical center.
Pre-assignment Details: The enrolled patients were pretreated with Thymoglobulin and methylprednisolone induction followed by combination therapy with both sirolimus (Rapa) and tacrolimus (FK) for 6 months. At 6 months, those without rejection on protocol biopsy with good tolerance to both drugs were randomized either Rapa or FK monotherapy and followed up for 48 months.
Groups:
- Sirolimus Group: Patients treated with sirolimus monotherapy from 6 months after combination therapy
- Tacrolimus Group: Patients treated with tacrolimus monotherapy from 6 months after combination therapy
Period: Overall Study
Arm/Group | Sirolimus Group | Tacrolimus Group
Started | 15 | 16
Completed | 7 | 8
Not Completed | 8 | 8
Not completed — Drug intolerance | 8 | 8

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed using the patients who finished study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus Group | Tacrolimus Group | Total
Number analyzed (Participants) | 7 | 8 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 44.4 (13.1) | 45.0 (15.2) | 44.7 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Allograft Rejection
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Sirolimus Group | Tacrolimus Group
Number analyzed (Participants) | 7 | 8
participants | 0 | 0

2. Secondary Outcome: The Rate of Significant Drug-associated Complications.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Sirolimus Group | Tacrolimus Group
Number analyzed (Participants) | 7 | 8
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sirolimus Group | Tacrolimus Group
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes